CLINICAL TRIAL: NCT04204018
Title: Measuring Practice Pattern Changes and Clinical Utility of a Novel Test for Preeclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qure Healthcare, LLC (Industry)
Collaborators: Progenity, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 01PRO2019
Record Dates: First submitted 2019-11-15; First posted 2019-12-18 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: The study will enroll practicing OB/GYNs in the US. All eligible and consented participants will complete 4 patient simulations. The intervention arm only will receive educational material about Progenity's test prior to these simulations, and be provided simulated Progenity test results in the simulated cases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental-arm providers will complete four simulated patient cases (CPVs) with two additions described in the next column:
  Interventions: Other: Experimental Arm
- Control (No Intervention): These providers will complete four simulated patient cases (CPVs) only.

INTERVENTIONS:
Other: Experimental Arm — * First, these providers will receive educational materials (e.g. a slide deck) meant to mimic what physicians will receive in the real-world market as they learn about the Progenity technology.
  * Second, within each of their four cases, intervention-arm physicians only will receive simulated test results from the Progenity PE test at the clinically-appropriate point in each case.
  Arms: Experimental

SUMMARY:
This study will collect high-quality data on how practicing obstetricians across the U.S. currently manage patients showing signs and/or symptoms of preeclampsia and how the results of Progenity's test change clinical decision making. To do so, this study leverages simulated patient cases called Clinical Performance and Value vignettes (CPVs) in a proven methodology to rapidly measure physician care decisions.

DETAILED DESCRIPTION:
This study will collect high-quality data on how practicing obstetricians across the U.S. currently manage patients showing signs and/or symptoms of preeclampsia and how the results of Progenity's test change clinical decision making. Data from this study will better illuminate the clinical use cases with the most significant impact on clinical decision making (and thus the largest potential clinical utility) and the associated physician characteristics (e.g., age, practice setting, training) associated with test adoption.

This study leverages simulated patient cases called Clinical Performance and Value vignettes (CPVs) in a proven methodology to rapidly measure physician care decisions. CPVs are a unique and scalable tool that standardizes practice measurement by having all providers care for the same (virtual) patients. With all providers caring for the same patients, the CPVs generate unbiased data that yields powerful insights into clinical decision making and how these decisions change with the introduction of a new product or solution. Data from the CPVs can quickly demonstrate the clinical utility of a solution, be published in peer-reviewed literature, inform marketing strategies and positively impact coverage and reimbursement decisions.

The study is a prospective cohort trial with five steps:

1. Enrollment: The study will enroll 110 practicing obstetrician/gynecologists (OB/GYNs) in the U.S. who are determined to be eligible by an eligibility screener.
2. Provider survey: Once providers are enrolled in the study, they will be asked to complete a questionnaire describing their practice and professional background.
3. Randomization: The 110 OB/GYNs will be randomized into equally-sized (55) control and intervention arms.
4. Education: The intervention-arm OB/GYNs will receive educational materials duplicating what physicians would receive in the real-world market as they adopt the Progenity technology. These materials are comprised of a slide deck and/or a fact sheet.
5. CPVs: Physicians will then complete the four CPV patient simulations in random order. Cases will be identical across the intervention and control arms, except that the intervention arm will receive Progenity PE test results at an appropriate point in each simulated case. All cases are presented on an online platform, participants are provided with unique weblinks, accessible via any internet-connected computer.

ELIGIBILITY:
Inclusion Criteria:

1. Board-certified in obstetrics/gynecology
2. Averaging at least 20 hours per week of clinical duties over the last six months
3. English speaking
4. Access to the internet
5. Informed, signed and voluntarily consented to be in the study

Exclusion Criteria:

1. Not board certified in obstetrics/gynecology at least 2 years prior
2. Averaging less than 20 hours per week of clinical duties over the last six months
3. Non-English speaking
4. Unable to access the internet
5. Do not voluntarily consent to be in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
CPV-measured cost difference | One week
  Difference in cost of suspected PE-related care between control and intervention physicians. (Cost is calculated by measuring differential rates of medical interventions/levels of care selected by each arm on their CPVs, and multiplying by Medicare reimbursement rates for these interventions/levels of care.)
CPV-measured clinical score difference | One week
  Difference in the overall, and the diagnostic and treatment quality scores between control and intervention physicians. Diagnostic and treatment scores are calculated as the percent correct on CPVs, and the overall score is a average score of the subcategory scores (percent correct).

SECONDARY OUTCOMES:
CPV-measured cost differences by use case | One week
  Difference in cost of suspected PE-related care between control and intervention physicians. (Cost is calculated by measuring differential rates of medical interventions/levels of care selected by each arm on their CPVs, and multiplying by Medicare reimbursement rates for these interventions/levels of care.) This will be examined for each of the four use cases to determine in which case(s) cost metrics most improved.
CPV-measured clinical score differences by use case | One week
  Difference in the overall, and the diagnostic and treatment quality scores between control and intervention physicians. Diagnostic and treatment scores are calculated as the percent correct on CPVs, and the overall score is a average score of the subcategory scores (percent correct). This will be examined for each of the four use cases to determine in which case(s) CPV scores most improved.
CPV-calculated baseline variation | One week
  Baseline (control physicians) levels of variation in the work-up and management of suspected PE patients. Variation is examined by looking at the range and standard deviation of the overall baseline scores for each CPV.

CONTACTS AND LOCATIONS:
Overall Officials: John Peabody, MD PhD, Principal Investigator — President, QURE Healthcare
Locations (1):
- QURE Healthcare, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Background] Peabody JW, Luck J, Glassman P, Jain S, Hansen J, Spell M, Lee M. Measuring the quality of physician practice by using clinical vignettes: a prospective validation study. Ann Intern Med. 2004 Nov 16;141(10):771-80. doi: 10.7326/0003-4819-141-10-200411160-00008. PMID 15545677
- [Background] Peabody JW, Strand V, Shimkhada R, Lee R, Chernoff D. Impact of rheumatoid arthritis disease activity test on clinical practice. PLoS One. 2013 May 7;8(5):e63215. doi: 10.1371/journal.pone.0063215. Print 2013. PMID 23667587
- [Background] Peabody J, Martin M, DeMaria L, Florentino J, Paculdo D, Paul M, Vanzo R, Wassman ER, Burgon T. Clinical Utility of a Comprehensive, Whole Genome CMA Testing Platform in Pediatrics: A Prospective Randomized Controlled Trial of Simulated Patients in Physician Practices. PLoS One. 2016 Dec 30;11(12):e0169064. doi: 10.1371/journal.pone.0169064. eCollection 2016. PMID 28036350
- [Background] Solon O, Woo K, Quimbo SA, Shimkhada R, Florentino J, Peabody JW. A novel method for measuring health care system performance: experience from QIDS in the Philippines. Health Policy Plan. 2009 May;24(3):167-74. doi: 10.1093/heapol/czp003. Epub 2009 Feb 18. PMID 19224955